CLINICAL TRIAL: NCT00987428
Title: Randomised Multicenter Trial of Early EUS Followed by Endoscopic Sphincterotomy in Case of Bile Duct Stone vs Conservative Treatment in Severe Biliary Pancreatitis
Brief Title: Early Endoscopic Ultrasound - Based Sphincterotomy or Conservative Treatment in Severe Biliary Pancreatitis
Acronym: EEPAB2
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Insufficient number of participants
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Collaborators: URC-CIC Paris Descartes Necker Cochin (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: P080903
Record Dates: First submitted 2009-09-29; First posted 2009-10-01 (Estimated); Last update posted 2025-11-20 (Actual); Status verified 2025-09

CONDITIONS: Pancreatitis Acute Biliary
Keywords: ERCP; EUS; Pancreatitis biliary; Severe; Interventional endoscopy; Choledocolithiasis
MeSH Terms: conditions — Lymphoma, Follicular | interventions — High-Energy Shock Waves

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- groupe 1 (Experimental): Early endoscopic ultrasonography and endoscopic sphincterotomy in case of common bile duct stone
  Interventions: Procedure: ultrasonography with or not sphincterotomy
- Groupe 2 (Active Comparator): usual procedure
  Interventions: Procedure: Usual procedure

INTERVENTIONS:
Procedure: ultrasonography with or not sphincterotomy — Early endoscopic ultrasonography and endoscopic sphincterotomy in case of common bile duct stone
  Arms: groupe 1
Procedure: Usual procedure — The control group includes patients with predicted severe ABP undergoing conservative treatment or endoscopic sphincterotomy (without EUS) within 72 hours of the onset of symptoms in case of cholangitis or biliary obstruction.
  Arms: Groupe 2

SUMMARY:
The primary purpose of this trial is to determine whether an early Early Endoscopic Ultrasound (EUS) immediately followed by an endoscopic sphincterotomy (ES) in case of bile duct stones may improve outcomes in patients with predicted severe acute biliary pancreatitis (ABP).

DETAILED DESCRIPTION:
The management of Acute biliary pancreatitis (ABP) remains controversial. Although early decompression of the bile duct is deemed potentially beneficial, previous randomised studies failed to show the benefit of early endoscopic sphincterotomy (ES) except in selected cases. However, those studies did not use recent non invasive diagnostic methods such as EUS.

Methodology: Patients in the study group undergo EUS followed by ES in case of common bile duct stones within 48 hours of the onset pf symptoms; The control group includes patients with predicted severe ABP undergoing conservative treatment or endoscopic sphincterotomy (without EUS) within 72 hours of the onset of symptoms in case of cholangitis or biliary obstruction.

ELIGIBILITY:
Inclusion criteria :

* age > 18
* predicted severe acute biliary pancreatitis (including age > 80, BMI >30, pre-existing organ failure, Modified Glasgow score > 3)
* timespan between onset and randomization < 48 hrs
* informed consent signed by patient or liable person in case of emergency

Exclusion criteria :

* non biliary pancreatitis
* non severe pancreatitis
* age < 18
* timespan between onset and randomization > 48 hrs
* absence of consent
* ongoing pregnancy
* no social security insurance

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 27 (Actual)
Dates: Start 2009-08; Primary Completion 2011-06 (Actual); Study Completion 2012-03 (Actual)

PRIMARY OUTCOMES:
The difference between the SOFA score measured at entry in the study (day 0) and at day 8 | Day 8

SECONDARY OUTCOMES:
Differences in SOFA score as measured at entry in the study and at day 15 | Day 15
Procedure-related morbidity | at Day 15 to 3 months
Overall morbidity | at day 15
Overall mortality | at day 15
Difference in Balthazar's scores (CT-scan) at entry and at days 8 and 15 | at day 8 and day 15

CONTACTS AND LOCATIONS:
Overall Officials: Frederic Prat, MD, PhD, Principal Investigator — Assistance Publique - Hôpitaux de Paris
Locations (1):
- Hopital Cochin, Paris, France